CLINICAL TRIAL: NCT01662544
Title: Comparison of Heated Humidified High-flow Nasal Cannula (HHFNC) Versus Standard Nasal Cannula Oxygen Delivery on Respiratory Distress and Length of Stay in Infants With Bronchiolitis and Hypoxia
Brief Title: Heated High Flow Oxygen Use in Infants With Bronchiolitis and Hypoxia
Acronym: HHFNC
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Children's Hospitals and Clinics of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1103-041
Record Dates: First submitted 2012-08-08; First posted 2012-08-10 (Estimated); Last update posted 2017-07-19 (Actual); Status verified 2017-07

CONDITIONS: Bronchiolitis; Hypoxia
Keywords: Infants; Bronchiolitis; Hypoxia; Emergency Department; Length of Stay; Pediatrics
MeSH Terms: conditions — Bronchiolitis; Hypoxia; Emergencies

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- HHFNC (Experimental): Heated High Flow arm
  Interventions: Procedure: Oxygen delivery
- Standard Nasal Cannula (Active Comparator): Standard treatment
  Interventions: Procedure: Oxygen delivery

INTERVENTIONS:
Procedure: Oxygen delivery

SUMMARY:
Bronchiolitis is a common cold weather seasonal respiratory illness affecting infants and children. Multiple supportive therapies have been tried in infants with bronchiolitis including albuterol, racemic epinephrine, hypertonic saline nebulization, but to date supportive therapy with oxygen is the only proven therapy to decrease respiratory distress in infants with bronchiolitis, with hypertonic saline showing a borderline statistically significant improvement. This prospective, randomized study will compare CSS and PEWS scores on infants who receive oxygen by standard flow nasal cannula and to those who receive oxygen via Humidified High-Flow Nasal Cannula (HHFNC). The results will help determine if infants with viral bronchiolitis who receive humidified high flow nasal cannula oxygen therapy have improved Clinical Severity Score (CSS) and Pediatric Early Warning System (PEWS) scores and ultimately decreased lengths of admissions when compared to patients treated with nasal cannula oxygen therapy with/without bronchodilator therapy.

Hypothesis Heated Humidified High-flow Nasal Cannula Delivery of Oxygen decreases respiratory distress as measured by pediatric CSS and PEWS when compared with routine nasal cannula oxygen delivery in infants with bronchiolitis.

ELIGIBILITY:
Inclusion Criteria:

1. Are previously healthy infants ages 3 months to 18 months of age
2. Have O2 saturations of < 92% on room air while awake
3. Have a clinical diagnosis of bronchiolitis
4. Have a CSS score showing moderate distress >4
5. Have a planned admission to the hospital for either inpatient or observation status
6. Have parental consent to enroll in study

Exclusion Criteria:

1. Have significant apnea or bradycardia events reported by parent or witnessed in Emergency Department
2. Have prior airway disease diagnosis other than URI within the previous two months
3. Were previously intubated; previously having had airway bronchoscopy or surgery
4. They are ex-preemies, i.e. had an estimated gestational age of <37 weeks at time of birth
5. Have a diagnosis of lobar consolidation or round pneumonia by Chest x-ray
6. Have pleural disease by chest x-ray
7. Have history of cardiac disease, renal disease, hematologic disease such as sickle cell disease or leukemia, congenital hemoglobinopathies or Congenital Adrenal Hyperplasia
8. Have undergone prior radiation or chemotherapy
9. Have functional or anatomical bowel obstruction as demonstrated by persistent vomiting or tensely distended abdomen
10. Have history of Choanal atresia or cleft palate
11. Have history of neuromuscular disorder, e.g., Spinal muscular atrophy, muscular dystrophies, cerebral palsy or hypotonia
12. Have impending respiratory failure as demonstrated by blood gas with pCO2 of greater than 60 or apnea spells lasting greater than 30 seconds

Ages: 3 Months to 18 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 56 (Actual)
Dates: Start 2012-08; Primary Completion 2015-05 (Actual); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
CSS Scores | Study specific

SECONDARY OUTCOMES:
PEWS Score | Study specific

OTHER OUTCOMES:
Oxygen needs | Study specific

CONTACTS AND LOCATIONS:
Overall Officials: Donna Milner, MD, Principal Investigator — Children's Hospitals and Clinics of Minnesota
Locations (1):
- Children's Hospitals and Clinics of Minnesota, Minneapolis, Minnesota, United States